CLINICAL TRIAL: NCT03013127
Title: PROMO: A Phase II Study of Pembrolizumab in Patients With Relapsed Or Metastatic Osteosarcoma Not Eligible for Curative Surgery
Brief Title: A Study of Pembrolizumab in Patients With Relapsed Or Metastatic Osteosarcoma Not Eligible for Curative Surgery
Acronym: PROMO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion of patients was stopped because ≤2 patients had clinical benefit.
Sponsor: Oslo University Hospital (Other)
Collaborators: Italian Sarcoma Group (Network); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kjetil Boye, MD PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK3475-482
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Osteosarcoma
Keywords: Osteogenic Sarcoma; Osteosarcoma; Sarcoma, Osteogenic; Pembrolizumab; Immunotherapy
MeSH Terms: conditions — Osteosarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab (MK-3475) 200 mg i.v. every 3 weeks for up to 35 cycles
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a humanized antibody used in cancer immunotherapy.
  Other Names: Keytruda

SUMMARY:
This is a phase II, single arm, open-label, interventional trial of pembrolizumab (MK-3475) in patients with osteosarcoma who have experienced disease relapse or progression after at least one line of systemic treatment, and who are not eligible for curative surgery.

DETAILED DESCRIPTION:
Patients with osteosarcoma, who are not eligible for surgery of curative intent and have completed at least one line of systemic therapy, will be considered for treatment with pembrolizumab. Patients who are considered medically unfit for chemotherapy and where no other treatment options are believed to be of major benefit may also be considered. Patients will receive pembrolizumab for up to 35 cycles.

Patients, who have received 35 cycles of pembrolizumab or discontinued study treatment of another reason than progression, will in the follow-up period be assessed for safety and treatment-related toxicity (for up to 90 days), progression and survival.

Patients who have achieved a clinically meaningful response after 35 cycles of pembrolizumab, defined as complete response (CR), partial response (PR), and stable disease (SD) assessed by the Investigator by using RECIST, v1.1, and have not experienced any clinically significant toxicity of study treatment, may be considered for reintroduction of pembrolizumab, if progression is detected > 8 weeks after cycle 35.

Due to the low incidence of osteosarcoma, the inclusion rate is expected to be low, thus a Simon's two-stage design is suggested. Evaluation of efficacy and safety in stage one will be performed after the first 12 patients have been treated for 18 weeks:

* In case of ≤2 responders; the trial ends.
* If ≥3 responders, the trial will continue into stage II to a total number of 25 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed osteosarcoma.
2. Disease relapse or progression after at least one line of systemic treatment.

   1. First-line systemic treatment should include cytotoxic chemotherapy according to local practice.
   2. The patient can be eligible if he/she is considered medically unfit for chemotherapy, as assessed by the sarcoma centre in charge of the patient's treatment.
3. Surgical resection with curative intent not possible.
4. Be willing and able to provide written informed consent/assent for the trial.
5. Be >18 years of age on day of signing informed consent.
6. Have measurable disease based on RECIST, version 1.1.
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen.
8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
9. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or sarcomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include sarcomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | At 18 weeks
  The percentage of patients with unresectable osteosarcoma who have achieved clinical response; complete response (CR), partial response (PR), or stable disease (SD) at 18 weeks as assessed using RECIST v1.1.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Assessments every 6-9 weeks up to 2 years
  The percentage of patients with unresectable osteosarcoma who have achieved objective response during treatment; complete response (CR), partial response (PR), as assessed using RECIST v1.1.
Progression-free survival (PFS) | Up to 4 years
Response rate by immune-related Response Criteria (ir-RC) | Assessments every 6-9 weeks up to 2 years
Overall survival (OS) | Through study completion, up to 4 years after enrollment of last patient
Number and type of Adverse Events related to pembrolizumab treatment in osteosarcoma patients as assessed by CTCAE v4.0 | Assessments every 6-9 weeks up to 2 years
  To evaluate the safety and tolerability of pembrolizumab in patients with osteosarcoma.
Health-related quality of life changes using EORTC QLQ-C30 | Assessments every 6-9 weeks up to 4 years
  To evaluate health-related quality of life changes from baseline in patients with osteosarcoma, receiving pembrolizumab, using EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Boye, MD, Principal Investigator — Oslo University Hospital
Locations (2):
- Istituto Ortopedico Rizzoli, Bologna, Italy
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boye K, Longhi A, Guren T, Lorenz S, Naess S, Pierini M, Taksdal I, Lobmaier I, Cesari M, Paioli A, Londalen AM, Setola E, Hompland I, Meza-Zepeda LA, Sundby Hall K, Palmerini E. Pembrolizumab in advanced osteosarcoma: results of a single-arm, open-label, phase 2 trial. Cancer Immunol Immunother. 2021 Sep;70(9):2617-2624. doi: 10.1007/s00262-021-02876-w. Epub 2021 Feb 12. PMID 33580363